CLINICAL TRIAL: NCT05403840
Title: Comparative STudy chaRacterising the Physiological changEs Induced by Surgical and tranScatheter Mitral Regurgitation Reduction (STRESS-MR)
Brief Title: Haemodynamics of Mitral Regurgitation Reduction
Acronym: STRESS-MR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Omar Chehab, Co-investigator, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: 1.4
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MVRR: Patients due to undergo surgical MV repair/replacement
  Interventions: Procedure: Mitral valve surgery
- TMVI: Patients due to undergo transcatheter MV intervention
  Interventions: Procedure: Transcatheter mitral valve intervention

INTERVENTIONS:
Procedure: Mitral valve surgery — Surgical mitral valve repair or replacement
  Groups: MVRR: Patients due to undergo surgical MV repair/replacement
Procedure: Transcatheter mitral valve intervention — Transcatheter mitral valve repair or replacement
  Groups: TMVI: Patients due to undergo transcatheter MV intervention

SUMMARY:
There is uncertainty in terms of the superiority of conventional valve surgery or percutaneous transcatheter intervention for the treatment of severe mitral regurgitation (MR) in high risk patients. The post procedural haemodynamics of the different treatment options in those at high surgical risk is poorly understood. This study seeks to characterise the physiological changes and functional outcomes of patients undergoing either surgery or transcatheter intervention.

DETAILED DESCRIPTION:
Conventional surgery for mitral regurgitation (MR) in high risk patients is associated with reduced benefit and increased risk of perioperative complications.Percutaneous transcatheter intervention (edge to edge repair) is an alternative treatment option is associated with clinical benefit and reduced peri-procedural risk. The post procedural haemodynamics of the different treatment options in those at high surgical risk is poorly understood.

This is a a prospective observational study, involving patients with severe MR undergoing mitral valve surgery (MVRR) and transcatheter intervention (TMVI) as standard of care being recruited into two separate cohorts. Patients will undergo investigations at baseline, in hospital post-operative, and at 6 months to characterise cardiac structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral regurgitation as per European Society of Cardiology guidelines
* Patients undergoing MVRR or TMVI as standard of care
* Patients at high, prohibitive surgical risk as judged by the Heart Team

Exclusion Criteria:

* Pregnancy and patients under the age of 18 years
* Congenital heart disease
* Moderate or severe mitral stenosis, aortic, pulmonary valve disease
* Patients currently enrolled in any other study where involvement in this study would involve deviation from either protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic severe mitral regurgitation accepted for either surgery or transcatheter valve intervention as standard of care and judged to be at high or prohibitive surgical risk.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-06 (Estimated); Primary Completion 2024-06-06 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular efficiency as measured by ventricular arterial coupling | From baseline to immediately following intervention and 6 months follow up
  VA coupling is calculated by the ratio of effective arterial elastance (Ea), a measure of afterload, to LV end systolic elastance (Ees), a relatively load independent measure of LV chamber performance. Both these measures are expressed in mmHg/ml and as continuous variables. Normal determined Ea and Ees values in resting subjects are 2.2 ± 0.8 mmHg/ml and 2.3 ± 1.0 mmHg/ml, respectively. When Ea/Ees ratio is approximately equal to 1.0, LV and arterial system are optimally coupled to produce stroke work, a measure of the efficiency of LV work, corresponding to the product of systolic arterial pressure and stroke volume, and related to oxygen consumption. When Ea/Ees ratio is <1.0, the stroke work remains close to optimal values, but when EA/EES ratio is >1.0, the stroke work significantly falls, and the LV becomes progressively less efficient. We will compare VA coupling before and after intervention and will be analyzed as continuous variables with appropriate statistical tests.

SECONDARY OUTCOMES:
Change in Left Ventricular End Diastolic Volume (LVEDV) | Baseline to 6 months post intervention
  Paired data comparing the Change in LVEDV at baseline vs 6 months
Change in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP Levels) | From baseline to immediately following intervention and 6 months follow up
Residual Mitral Regurgitation (MR) Severity | Immediately following intervention and 6 months follow up
  MR Severity Grading done by Quantitative Doppler Echocardiography
Change in New York Heart Association (NYHA) Functional Class | Baseline to 6 months follow up
  The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity:
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms Class IV - Severe limitations.
Change in Six Minute Walk Test (6MWT Distance or 6MWD) | Baseline to 6 months follow up
  The Six Minute Walk Test (6MWT) is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk ona flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation,peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity.
Change in Quality of Life (QoL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to 6 months follow up
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score. Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification. Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.

IPD SHARING:
Plan to Share IPD: No
To be determined.